CLINICAL TRIAL: NCT02467946
Title: A Phase 1/2 Clinical Trial to Assess Safety and Efficacy of a New Treatment for Hodgkin Lymphoma's Disease Combining Adcetris® and Levact® in Old Patients
Brief Title: Hodgkin Lymphoma Treatment With Adcetris and Levact in the Old Patient
Acronym: HALO
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centre Antoine Lacassagne (Other)
Collaborators: Millennium: The Takeda Oncology Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013/24
Record Dates: First submitted 2015-06-04; First posted 2015-06-10 (Estimated); Last update posted 2023-01-04 (Actual); Status verified 2022-04

CONDITIONS: Clinical Efficacy; Safety
MeSH Terms: interventions — Bendamustine Hydrochloride; Brentuximab Vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Adcetris-Levact (BV-Be) Association (Experimental): Adcetris® (BV) : 1.2 mg/kg intravenously every 3 weeks Levact® (Be): 90 mg/m2/day intravenously for 2 days every 3 weeks. Up to 6 cycles
  Interventions: Drug: Adcetris-Levact

INTERVENTIONS:
Drug: Adcetris-Levact — Association of Adcetris (1.2 mg/kg intravenously every 3 weeks) with Levact (90 mg/m2/day intravenously for 2 days every 3 weeks) during at least 6 cycles.
  Other Names: Bendamustine; Brentuximab Vedotin

SUMMARY:
Treatment outcome with ABVD in elderly patients remains inferior to adults. Moreover, Bleomycin-induced lung toxicity in the elderly has been reported as high as 46%. For these reasons, questions arise whether ABVD could be still considered the standard treatment in HL patients aged > than 60. Regimens containing other alkylators such as CHOP proved even superior to ABVD, with a 3-y PFS of 67%. Frontline treatment of advanced-stage HL with Brentuximab Vedotin (BV) in association with AVD (Doxorubicin, Vinblastine, Dacarbazine) proved very active in a pioneer study, reporting the preliminary results of a phase 1 multicentre trial, in which the percentage of patients achieving CR was as high as 92%. For all these reason the investigators decided to test the association of an alkylator with an innovative mechanism of action and a very safe toxicity profile in the elderly such as Bendamustine (Be) with BV in untreated elderly HL patients.

The combination of BV and Be, investigated in this study, might represent an innovative treatment alternative for HL patients older than 60 years of age, especially for those of them in whom ABVD chemotherapy, the current standard front-line treatment, is not suitable. However, even when ABVD is given as upfront treatment for elderly HL patients, it is associated with substantial dose reduction, treatment delay, toxicity, and treatment-related mortality, with treatment outcomes remaining much inferior to those obtained in younger patients. This drug association is expected to be safe, well-tolerated and to demonstrate higher efficiency compared with ABVD. In this setting, it is expected that this therapy could be offered to the large majority of elderly patients with a full treatment completion reached in up to 80% of these patients.

Thus, the aim of this study will be to assess safety and efficacy of the above association.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with advanced classical Hodgkin Lymphoma according to the World Health Organization classification. All Hasenclever IPS prognostic groups accepted
2. Stages IIB to IV B
3. Age 60-80 years included
4. Patient not previously treated
5. ECOG ≤ 2
6. Patient with adequate organ function:

   * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
   * Haemoglobin ≥ 9 g/dL
   * Platelets (PTL) ≥ 100 x 109/L
   * AST - ALAT ≤ 2.5x ULN
   * Bilirubin ≤ 1.5 x ULN
   * Creatinine < 150 µmol/l (or 1.7 mg/dl)
7. Male patients, even if surgically sterilized, (i.e., status post vasectomy) and women of childbearing potential agree to practice effective barrier contraception during the entire study period and through 6 months after the last dose of study drug, or agrees to completely abstain from heterosexual intercourse.

   • Contraception as described above is not a requirement if the female patient's postmenopausal status is documented (has had no menstrual period for at least 12 consecutive months)
8. Information delivered to patient and voluntary written informed consent must be given before performance of any study-related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.
9. Patient affiliated with a health insurance system.

Exclusion Criteria:

1. Patients aged less than 60 years.
2. Diagnosed or treated for another malignancy within 3 years before the first dose or previously diagnosed with another malignancy and have evidence of residual disease. Patients with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
3. Known cerebral or meningeal disease (HL or any other etiology), including signs or symptoms of PML.
4. Symptomatic neurologic disease compromising instrumental activities of daily living or requiring medication.
5. Symptomatic sensory or motor peripheral neuropathy.
6. Concurrent use of other investigational agents. In case of previous participation to a Clinical trial, a period of 30 days will be observed after the end of the previous Clinical Trial and before the inclusion in HALO study
7. Chemotherapy, biologics, and/or other treatment with immunotherapy not completed at least 4 weeks prior to first dose of study drug.
8. Patient who had major surgery less than 30 days before start of treatment
9. Any active systemic viral, bacterial, or fungal infection requiring systemic antibiotics within 2 weeks prior to first study drug dose.
10. Known hypersensitivity to recombinant proteins, murine proteins, or to any excipient contained in the drug formulation of BV.
11. Patient presenting an uncontrolled infectious disease, including active HBV infection defined by either detection of HBs Antigen or presence of anti HBc antibody without detectable anti HBs antibody or HIV or HCV serology positivity. In case of HBc positive serology, a PCR could be performed in order to determine viral load. Patients with viral load defined as negative could be included.

    o A prophylactic treatment will be strongly recommended (see HALO Study protocol, paragraph 6.2.3, page 36)
12. Patient with history of poor compliance or current or past psychiatric conditions or severe acute or chronic medical conditions, or laboratory abnormalities that would interfere, in the judgment of the investigator and/or sponsor, with the ability to comply with the study protocol.
13. Patients with uncompensated diabetes mellitus and fasting glucose levels over 180 mg/dl.
14. Known history of any of the following cardiovascular conditions

    * Myocardial infarction within 2 years of enrollment
    * New York Heart Association (NYHA) Class III or IV heart failure (see Appendix 12)
    * Evidence of current uncontrolled cardiovascular conditions, including cardiac arrhythmias, congestive heart failure (CHF), angina, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities
15. Recent evidence (within 6 months before first dose of study drug) of a left-ventricular ejection fraction <50%
16. People particularly vulnerable including:

    * Person deprived of liberty
    * Adult patient entitled to protection of law

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-01-14 (Actual); Primary Completion 2022-04-06 (Actual); Study Completion 2022-04-06 (Actual)

PRIMARY OUTCOMES:
toxicity analysis | up to 2.5 years
  To evaluate the tolerability and toxicity of Adcetris-Levact (BV-Be) association.
Efficacy analysis | up to 2.5 years
  To evaluate the efficacy in terms of Response Rate after treatment completion of Adcetris-Levact (BV-Be) association.

SECONDARY OUTCOMES:
Progression Free Survival | 3 years
  * To evaluate the efficacy in terms of:
  * Progression Free Survival at 3 years
  * Event Free Survival at 3 years
  * Overall Survival at 3 years
Complete Response Rate | 2 years
  • To evaluate the efficacy in terms of Complete Response Rate after two cycles of Adcetris-Levact (BV-Be) association

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Antoine Lacassagne, Nice, France

REFERENCES:
- See also: Related Info — http://www.centreantoinelacassagne.org